CLINICAL TRIAL: NCT00985322
Title: A Prospective, Randomized, Open Label, Blinded End-point (Probe) Trial to Evaluate Whether, at Comparable Blood Pressure Control, ACE Inhibitor Therapy More Effectively Than Non RAS Inhibitor Therapy Reduces CArdiovascular Morbidity and Mortality in Chronic DIAlysis Patients With Left Ventricular Hypertrophy and/or Arterial Hypertension (ARCADIA Study)
Brief Title: Angiotensin-converting-enzyme (ACE) Inhibitors in Hemodialysis
Acronym: ARCADIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCADIA; 2008-003529-17 (EudraCT Number)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Left Ventricular Hypertrophy; Hypertension
Keywords: Hemodialysis
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE inhibitor Ramipril (Experimental)
  Interventions: Drug: ACE inhibitor Ramipril
- non-RAS inhibitor antihypertensive therapy (Active Comparator)
  Interventions: Drug: non-RAS inhibitor antihypertensive therapy

INTERVENTIONS:
Drug: ACE inhibitor Ramipril — The ACE inhibitor (Ramipril) will be started at 1.25 mg/day and will be up-titrated to 2.5 mg/day, to 5 mg/day, and then to 10 mg/day according to BP control and tolerability.
  Arms: ACE inhibitor Ramipril
Drug: non-RAS inhibitor antihypertensive therapy — Blood Pressure lowering regimen not including RAS inhibitors
  Arms: non-RAS inhibitor antihypertensive therapy

SUMMARY:
Background: Angiotensin-converting-enzyme (ACE) inhibitors have a specific cardioprotective effect and, compared to treatment not directly interfering with the renin-angiotensin-system (RAS), significantly reduce cardiovascular (CV) mortality and morbidity in subjects with normal renal function.

Despite CV events are the leading cause of death in these patients, no adequately powered trial so far evaluated the specific cardioprotective effect of ACE inhibitors in this population.

Objectives: This prospective, randomized, open label, blinded end point (PROBE) trial is primarily aimed at evaluating whether, at comparable blood pressure (BP) control, ACE inhibitor as compared to non-RAS inhibitor therapy significantly reduces the incidence of a composite end point of CV death (including sudden death) and non-fatal myocardial infarction or stroke in 266 patients with arterial hypertension (pre-dialysis systolic/diastolic BP >140/90 mmHg or post-dialysis systolic/diastolic BP >130/80 mmHg or antihypertensive therapy) and/or echocardiography evidence of LVH (cardiac mass index >130 g/m2 for men and 100 g/m2 for women) who are on dialysis therapy since at least six months. Secondarily, the study will compare the incidence of single components of the primary outcome, new onset paroxysmal or persistent atrial fibrillation, thrombosis of the artero-venous fistula, new onset, progression or regression of LVH, changes in components of the metabolic syndrome, the safety profile of the two treatment regimens and their cost/effectiveness.

Methods: After 1 month wash-out period from previous RAS inhibitor therapy and a baseline evaluation of main clinical and laboratory parameters, patients will be randomized on a 1:1 basis to 2-year treatment with an ACE inhibitor or a BP lowering regiment not including RAS inhibitors. A balanced distribution according to centre, number of dialysis sessions per week (2 or 3), presence of diabetes (YES/NO), arterial hypertension (YES/NO), LVH (YES/NO) will be achieved by the minimization method. Treatment will be adjusted to achieve and maintain a target BP <140/90 mmHg (pre-dialysis) and a target BP <130/80 mmHg (post-dialysis) in both groups.

Expected results: ACE inhibitor compared to non-RAS inhibitor therapy is expected to reduce more effectively fatal and non-fatal CV events, prevent or limit progression or induce regression of LVH, improve some components of the metabolic syndrome, and reduce treatment costs for cardiovascular complications. These findings might help achieving more effective cardioprotection in people on chronic dialysis at lower costs.

DETAILED DESCRIPTION:
Angiotensin converting enzyme (ACE) inhibitors have the broader effect of any drug in cardiovascular medicine, reducing the risk of death, myocardial infarction, stroke, diabetes, and renal impairment.A recent meta-analysis of 33,500 patients included in six randomized clinical trials and a pooled analysis of the Heart Outcomes Prevention Evaluation (HOPE), the European Trial on Reduction of Cardiac Events with Perindopril in Stable Coronary Artery Disease (EUROPA, and the Prevention of Events with Angiotensin-Converting-Enzyme Inhibition (PEACE) trials showed that ACE inhibitors reduce mortality and cardiovascular events also in subjects with coronary artery disease but preserved left ventricular function. However, all the above studies excluded patients with advanced renal insufficiency or end stage renal disease (ESRD). Thus, whether ACE inhibitors may have a specific cardioprotective effect also in this typology of patients is still matter of investigation. This is an issue of major clinical relevance since CV disease is the primary cause of morbidity and mortality in the ESRD population and affects as many as 50-60% of ESRD patients.The burden of CV disease in this population is predicted to dramatically increase over the next few years because of the rapidly increasing number of patients requiring renal replacement therapy and the increasing prevalence of ESRD patients at increased cardiovascular risk because of older age, diabetes and hypertension.

Despite the excess CV risk, a consistent proportion of ESRD patients are not given ACE inhibitor therapy because of concern of hyperkalemia. Others, on the contrary, are treated on the basis of results of available trials. However, whether data in subjects without renal insufficiency can be generalized also to those with ESRD is unknown. This is an itchy point since dialysis patients might respond differently to therapies of proven benefits in non-ESRD patients. For instance, data from the German Diabetes and Dialysis study showed that, unlike in the general population, HmGCoA inhibitor therapy failed to decrease CV mortality in a hemodialysis population. Thus, ad hoc studies in the ESRD population are urgently needed. A recent trial, the Fosinopril in Dialysis (FOSIDIAL) study, tried to address this issue, but was clearly underpowered and results were inconclusive. However, evidence of a non significant trend to less cardiovascular events in the ACE inhibitor arm, suggests that ACE inhibitors might have a specific cardioprotective effect also in this population.

Thus, whether ACE inhibitor therapy more effectively than non-RAS inhibitor therapy reduces CV morbidity in high risk patients on chronic dialysis therapy is worth investigating in an adequately powered trial.

Aims

The broad aim of the study is to evaluate whether ACE inhibitor therapy reduces CV mortality and morbidity in high-risk ESRD patients with arterial hypertension and/or LVH who are on chronic hemodialysis therapy since >6 months.

Primary:

* To assess whether, at comparable BP control, ACE inhibitor as compared to non-RAS inhibitor therapy reduces the incidence of a combined end-point of CV death (including sudden cardiac death and cardiac arrest resuscitation) and myocardial infarction or non-fatal stroke.

Secondary:

* To compare the incidence of the single components of the combined end-point, of myocardial or peripheral revascularizations, new onset of atrial fibrillation in one of its three forms (paroxysmal, persistent and permanent) or recurrence of the arrhythmia in patients who experienced paroxysmal or persistent atrial fibrillation previously, hospitalizations for chronic heart failure and thrombosis of the artero-venous fistula.
* To evaluate whether ACE inhibitors prevent, limit progression or achieve regression of LVH and ameliorate some of the components of the metabolic syndrome and whether these effects correlates with CV outcomes.
* To compare the cost/effectiveness of the two treatments.

Safety:

* Serious (including disturbances of cardiac rhythm and electrical conduction possibly related to hyperkalemia) and non-serious adverse events.
* Any clinical or laboratory abnormality -such as symptomatic hypotension, cough, hyperkalemia (serum potassium >6 mEq/L), anemia requiring increasing doses of erythropoietin- possibly related to ACE inhibitor therapy.

Design:

This prospective, randomized, open label, blinded end point (PROBE) trial will include 266 hypertensive ESRD patients with echocardiography evidence of LVH who are on chronic hemodialysis since >6 months. After 1 month wash-out period from previous RAS inhibitor therapy and stratification for diabetes YES/NO, they will have a baseline evaluation of main clinical and laboratory parameters and will be randomized to 2-year treatment with an ACE inhibitor or a BP lowering regimen not including RAS inhibitors. Treatment will be adjusted to achieve and maintain a target BP <140/90 mmHg (pre-dialysis) and a target BP <130/80 mmHg (post-dialysis) in both groups.

ELIGIBILITY:
Inclusion criteria:

* Men and women >18 years of age who are on chronic renal replacement treatment since at least 6 months with two or three haemodialysis sessions per week.
* Hypertension (pre-dialysis systolic and/or diastolic BP >140/90 mmHg or post-dialysis systolic and/or diastolic BP >130/80 mmHg or ongoing antihypertensive therapy).

and/or

* LVH defined by a cardiac mass index >130 g/m2 for men and 100 g/m2 for women (17) within three months of enrolment.
* Written informed consent.

Exclusion criteria:

* Specific indication (such as heart failure) or contraindication (such as hypersensitivity) to ACE inhibitor therapy.
* Any concomitant medication with ACE inhibitors and angiotensin II receptor antagonists
* Hyperkalemia (serum potassium >6 mEq/L) despite optimal control of metabolic acidosis and blood glucose (in diabetics) in patient with less then three dialysis sessions per week.
* Symptomatic chronic or intradialytic hypotension.
* Arrhythmias that in the Investigator judgement might be worsened by hyperkalemia (such as sinus bradycardia, delayed atrio-ventricular conduction, atrio-ventricular blocks).
* CV events (stroke, acute myocardial infarction or other acute coronary syndromes) over the last three months.
* Uncontrolled hyper- or hypo-thyroidism.
* Active systemic disease, malignancies and any clinical condition associated with a life-expectancy of less than 2 years.
* Drug or alcohol abuse, psychiatric disorders and inability to understand the potential risks or benefits of the study.
* Pregnancy, lactation or child bearing potential and ineffective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2009-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The main outcome variable will be a combined end-point of cardiovascular death (including sudden death and cardiac arrest resuscitation) and myocardial infarction or non-fatal stroke. | Baseline, 1st and 2nd year

SECONDARY OUTCOMES:
Single components of combined endpoint,myocardial or peripheral revascularizations,new onset paroxysmal,persistent or permanent or recurrence of atrial fibrillation,hospitalizations for chronic heart failure,and thrombosis of artero-venous fistula | Baseline, 1st and 2nd year

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (29):
- Italy (29):
  - Policlinico San Pietro, Ponte San Pietro, Bergamo
  - Ospedale "Treviglio-Caravaggio", Treviglio, Bergamo
  - Hospital of Montichiari, Montichiari, Brescia
  - Presidio Ospedaliero Acireale, Acireale, Catania
  - Hospital "Morgagni-Pierantoni", Forlì, Forlì Cesena
  - A.O. Desio e Vimercate, Desio, MB
  - Ospedale "Caduti Bollatesi", Bollate, Milano
  - Hospital of Cernusco sul Naviglio, Cernusco sul Naviglio, Milano
  - Hospital "Bassini", Cinisello Balsamo, Milano
  - A.O. Ospedale Civile di Legnano, Legnano, Milano
  - A.O. della Provincia di Lodi, Lodi, Milano
  - Presidio Ospedaliero di Magenta, Magenta, Milano
  - IRCCS "Humanitas", Rozzano, Milano
  - IRCCS Multimedia, Sesto San Giovanni, Milano
  - Fondazione San Raffaele Monte Tabor, Milan, MI
  - Ospedale San Giovanni di Dio, Agrigento
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Hospital "Ospedali Riuniti ", Bergamo
  - Hospital "Policlinico S.Orsola-Malpighi", Bologna
  - A.O. Giuseppe Brotzu, Cagliari
  - ASL 8 - S.C. Territoriale di Nefrologia e Dialisi, Cagliari
  - A.O. S. Croce e Carle, Cuneo, Cuneo
  - Hospital "San Paolo", Milan
  - Hospital "San Gerardo", Monza
  - Hospital "Azienda Ospedaliera Universitaria Di Parma", Parma
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Hospital "Degli Infermi", Rimini
  - A.O. Umberto I, Syracuse
  - P.O. G. Mazzini, Teramo

REFERENCES:
- [Derived] Ruggenenti P, Podesta MA, Trillini M, Perna A, Peracchi T, Rubis N, Villa D, Martinetti D, Cortinovis M, Ondei P, Condemi CG, Guastoni CM, Meterangelis A, Granata A, Mambelli E, Pasquali S, Genovesi S, Pieruzzi F, Bertoli SV, Del Rosso G, Garozzo M, Rigotti A, Pozzi C, David S, Daidone G, Mingardi G, Mosconi G, Galfre A, Romei Longhena G, Pacitti A, Pani A, Hidalgo Godoy J, Anders HJ, Remuzzi G; ARCADIA Study Organization. Ramipril and Cardiovascular Outcomes in Patients on Maintenance Hemodialysis: The ARCADIA Multicenter Randomized Controlled Trial. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):575-587. doi: 10.2215/CJN.12940820. Epub 2021 Mar 29. PMID 33782036